CLINICAL TRIAL: NCT06268288
Title: Pilot Study--The Effects of Non-invasive Vagal Neurostimulation (nVNS) in Adolescents With Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Non-invasive Vagal Neurostimulation (nVNS) in Adolescents With Postural Orthostatic Tachycardia Syndrome (POTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lytitia M. Shea, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-011492
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome; Autonomic Dysfunction; Postural Orthostatic Tachycardia Syndrome; POTS - Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: Half of the patient population will be randomized to standard management only. The other half of the population will be randomized to standard management plus use of the vagal nerve stimulator
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS (Active Comparator): The General Pediatric and Adolescent Medicine providers at Mayo Clinic utilize a specific management program for their patients with Postural Orthostatic Tachycardia Syndrome utilizing the acronym STEPS. S is for liberal intake of salt, T is for drinking 90-100 ounces/day of fluid, E is for slowly and gradually improve continuous aerobic exercise duration to a goal of 50 minute most days of the week, P is for possible utilization of 1 of two prescription medications (metoprolol or midodrine), and S is for setting priorities and goals such as encouraging good sleep hygiene, attendance at school, social interactions, and counseling.
  Interventions: Other: STEPS management protocol
- STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation) (Experimental): Utilization of STEPS management goals plus the addition of non invasive vagal nerve stimulators for two 2 minutes of intervention performed three times a day.
  Interventions: Device: GammaCore intervention; Other: STEPS management protocol

INTERVENTIONS:
Device: GammaCore intervention — Use of the vagal nerve stimulator, GammaCore, on the right side of the neck for two 2 minute stimulations performed 3 times a day
  Other Names: external vagal nerve stimulator, non-invasive vagal nerve stimulator
  Arms: STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Other: STEPS management protocol — STEPS is the acronym for the standard management program for our patients with POTS. It includes liberal use of salt, taking in 90-100 ounces of fluid, gradually increasing the duration of aerobic exercise, possible use of one of two prescription medications (metoprolol, and midodrine), and encouragement to set priority and goals

SUMMARY:
The purpose of this study is to determine if nVNS will decrease autonomic symptom intensity (COMPASS-31 and Child Functional Disability Inventory) in adolescent patients with postural orthostatic tachycardia syndrome (POTS) in comparison to standard recovery STEPS management.

DETAILED DESCRIPTION:
Project purpose: The investigators will study the use of non invasive vagal nerve stimulation in newly diagnosed adolescent patients with POTS to see if symptom management improves over 2 months. Surveys will include COMPASS-31. Child Functional Disability Inventory, and PHQ-9. Patient logs will evaluate headache frequency, exercise duration and VNS use.

Research objectives: The investigators hypothesize that:

Primary Aim 1. Use of noninvasive vagal nerve stimulation will decrease autonomic symptom intensity compared to control group.

Primary Aim 2. Use of noninvasive vagal nerve stimulator will improve child function.

Primary Aim 3. Heart rate elevation measured by head up tilt table test will decrease in the treatment group compared to the control group.

Secondary goals include:

Secondary Aim 1: To determine if utilization of noninvasive vagal nerve stimulation influences headache frequency

Secondary Aim 2: Determine if utilization of noninvasive vagal nerve stimulation will influence weekly duration of aerobic exercise.

Secondary Aim 3: Determine if utilization of noninvasive vagal nerve stimulator results in significant side effects, particularly depression, in adolescent patients.

ELIGIBILITY:
Inclusion criteria:

1. Patient's age 12-19 years of age
2. Newly diagnosed POTS at Mayo Clinic in Rochester
3. Head up tilt table test results in a heart rate increase of 40 or more bpm
4. Consent is able to be obtained appropriately per age

Exclusion criteria:

1. POTS patients with orthostatic hypotension
2. POTS patients with vasovagal syncope
3. Use of medications other than midodrine or metoprolol
4. Inability to independently utilize the GammaCore device
5. Inability to independently complete surveys or patient logs
6. Patients receiving hormonal therapy other than birth control
7. Pregnancy
8. Prior neck surgery
9. Metallic implant present
10. Cardiac disorder
11. Presence of an eating disorder
12. Use of a feeding tube

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lytitia Shea, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS: The General Pediatric and Adolescent Medicine providers at Mayo Clinic utilized a specific management program for their patients with Postural Orthostatic Tachycardia Syndrome utilizing the acronym STEPS. S is for liberal intake of salt, T is for drinking 90-100 ounces/day of fluid, E is for slowly and gradually improve continuous aerobic exercise duration to a goal of 50 minute most days of the week, P is for possible utilization of 1 of two prescription medications (metoprolol or midodrine), and S is for setting priorities and goals such as encouraging good sleep hygiene, attendance at school, social interactions, and counseling.
  STEPS management protocol: STEPS is the acronym for the standard management program for our patients with POTS. It includes liberal use of salt, taking in 90-100 ounces of fluid, gradually increasing the duration of aerobic exercise, possible use of one of two prescription medications (metoprolol, and midodrine), and encouragement to set priority and goals
Period: Overall Study
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome Management/ STEPS | STEPS + GammaCore Intervention (Noninvasive Vagal Nerve Stimulation) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participants was limited to 12 years through 18 years of age
  years | 15 (3) | 16 (3) | 15 (3)
Sex: Female, Male [Count of Participants; unit: Participants] — Stratified randomization was used to ensure an equal number of males in the two arms of the studies. This was done to balance the few males expected in the study compared to females. Diagnoses of POTS in adolescents occurs primarily in females.
  Participants
    Female | 17 | 17 | 34
    Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Change in Composite Autonomic Symptom Score (COMPASS-31)
Description: The change in COMPASS-31 score from baseline to 8 weeks. COMPASS-31 measures autonomic dysfunction in patients with neurodegenerative diseases. It consists of 31 patient-reported questions assessing various symptoms, including orthostatic intolerance, vasomotor symptoms, and gastrointestinal issues. Total scores range from 0 to 100, with higher scores indicating more severe symptoms.
Time Frame: Baseline; 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 13 | 15
score on a scale | -5.40 (6.82) | -5.94 (10.89)

2. Primary Outcome: The Change in Child Functional Disability Inventory Scores
Description: The change in Child Functional Disability Inventory scores from baseline to eight weeks. The Child Functional Disability Inventory assesses the physical and psychosocial functioning of children due to their physical health. It consists of 15 items that measure activity limitations due to being sick or not feeling well. The total scores range from 0 to 60 with higher scores indicating greater perceived functional disability.
Time Frame: Baseline; 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 13 | 15
score on a scale | -2.92 (8.60) | -3.40 (11.76)

3. Primary Outcome: The Change in Heart Rate (Beats Per Minute) in Head up Tilt Table Tests
Description: The change in heart rate, measured in beats per minute (BPM), in the head up tilt table test (HUTT) from baseline to 8 weeks.
Time Frame: Baseline; 8 Weeks
Population: Everyone had a baseline head up tilt table test. The repeat tilt table test was voluntary and resulted in fewer patients participating in this repeat test. The reason we made this voluntary is that many participants live far away and return for a repeat head up tilt table is inconvenient and costly.
Measure: Mean (Standard Deviation); unit: Beats per Minute (BPM)
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 4 | 7
Beats per Minute (BPM)
  Baseline | 47.50 (6.45) | 58.14 (28.94)
  8 Weeks | 42.50 (7.00) | 40.14 (14.35)

4. Secondary Outcome: Change in the Number of Headaches Experienced by Adolescent Patients With POTS
Description: The change in the number of headaches from baseline to 8 weeks experienced by adolescent patients with POTS.
Time Frame: Baseline; 8 Weeks
Population: One patient in the standard POTS management/STEPS arm and two patients in the STEPS + GammaCore arm did not fill out the patient log at week 8 that documented the number of headaches they experienced. Due to this, no data exists for week 8 for these patients.
Measure: Median (Full Range); unit: Headaches
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 15 | 15
Headaches
  Baseline | 1.00 [1.00 to 2.10] | 1.30 [0.70 to 3.10]
  8 Weeks: number analyzed (Participants) | 14 | 13
  8 Weeks | 1.20 [0.60 to 2.00] | 0.40 [0.00 to 1.70]

5. Secondary Outcome: Change in Exercise Duration (Minutes) in Adolescent Patients With POTS
Description: The change in the exercise duration (minutes) in adolescent patients with POTS from baseline to 8 weeks.
Time Frame: Baseline; 8 Weeks
Population: One patient in the standard POTS management/STEPS arm and two patients in the STEPS + GammaCore arm did not fill out the patient log at week 8 that documented exercise duration in minutes. Due to this, no data exists for week 8 for these patients.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 15 | 15
Minutes
  Baseline | 25.00 [15.70 to 47.10] | 21.40 [8.60 to 45.70]
  8 Weeks: number analyzed (Participants) | 14 | 13
  8 Weeks | 32.50 [18.60 to 55.70] | 17.90 [10.00 to 45.00]

6. Secondary Outcome: Change in PHQ-9 Scores in Adolescent Patients With POTS
Description: The change in the Patient Health Questionnaire 9-item (PHQ-9) scale score from baseline to 8 weeks. PHQ-9 is used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
Time Frame: Baseline; 8 Weeks
Population: Seven patients in the Device group and seven patients in the Control group had incomplete data for the PHQ-9 scores (missing either the baseline PHQ-9 survey or the final PHQ-8 at 8 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
Number analyzed (Participants) | 13 | 13
score on a scale | 0.23 (3.56) | -3.39 (4.54)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 8 weeks.
Description: Adverse events were collected through patient logs and questionnaires.
Arm/Group | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Postural Orthostatic Tachycardia Syndrome management/ STEPS (N=20) | STEPS + GammaCore Intervention (noninvasive vagal nerve stimulation) (N=20)
Worsening Depression (Psychiatric disorders) | 0 | 1
Increase Headaches (Nervous system disorders) | 4 | 4
Increased Dizziness (Nervous system disorders) | 0 | 3
Bloating/Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Increased Anxiety (Psychiatric disorders) | 0 | 2
Loose Stool (Gastrointestinal disorders) | 1 | 0
Mood Swings (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT06268288/Prot_SAP_000.pdf